CLINICAL TRIAL: NCT02595151
Title: Real-time Observation of Microcirculatory Hemodynamics in Gastric Intestinal Metaplasia by Confocal Laser Endomicroscopy: a Feasibility Study
Brief Title: Real-time Observation of Microcirculatory Hemodynamics in Gastric Intestinal Metaplasia by Confocal Laser Endomicroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital, Shandong University
Other Study IDs: 2015SDU-QILU-G001
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-09

CONDITIONS: Flow Determination
Keywords: Probe-based confocal laser endomicroscopy; chronic atrophic antral gastritis; microcirculatory dynamics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Targeted fresh biopsy samples from each examined site were fixed in 10% pH neutral formalin, and embedded in paraffin. Slides of 4-um sections were deparaffinized and hydrated. After antigen retrieval and blocking procedures, Immunology and Histology Chemistry (IHC) staining for CD34 was performed by mouse anti-CD34 monoclonal antibody (ZM-0046, ZSGB-BIO, Beijjing, China) as per the manufacturers' instructions.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- gastric intestinal metaplasia: Those fulfilling the criteria of GIM by CLE according to the study by Yuting Guo et al were included.
  Interventions: Device: CLE
- normal gastric: diagnosed during routine colonoscopy procedures.
  Interventions: Device: CLE

INTERVENTIONS:
Device: CLE — The CLE procedure did not differ from that of conventional colonoscopy, except for the additional storage of pCLE images and videos in the gastric antrum.

SUMMARY:
The morphologic change of microvessels has the clinical value to distinguish cancerous from non-cancerous mucosa. The aim of this study was to observe gastric mucosa microcirculatory hemodynamic changes real-time using pCLE, compare the differences between chronic nonatrophic gastritis and GIM; then evaluate the possible mechanisms associated with gastric mucosal blood flow in GIM.

DETAILED DESCRIPTION:
Consecutive patients with GIM under endoscopic surveillance or examination at Qilu Hospital from March 1 to September 31, 2015 were recruited into this study. Before the endomicroscopic examination, 20,000 U α-chymotrypsin and 80 mg dimethylpolysiloxane were given orally to remove gastric mucus. All patients were given intravenous injections of 1 ml of 2% fluorescein sodium (Baiyunshan Mingxing Pharmaceutical, Guangzhou, China) as an allergy test before procedures were carried out. Conscious sedation was achieved for each patient by using propofol and fentanyl, and vital signs were monitored during the entire procedure. After successful intubation of the endoscope into the gastric antrum, 1 mL fluorescein sodium solution was applied intravenously as a contrast dye. The CLE procedure did not differ from that of conventional colonoscopy, except for the additional storage of pCLE images and videos in the gastric antrum. Finally, targeted biopsy of the examined site was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged 18-80 ;
2. Those fulfilling the criteria of GIM according to the study by Yuting Guo et al were included.

Exclusion Criteria:

1. patients younger than 18 years or older than 80 years;
2. finding of acute GI bleeding, gastrectomy or known upper gastrointestinal cancer;
3. unwillingness to participate in this study;
4. contraindications to CLE, such as fluorescein allergy, hepatic or renal dysfunction, jaundice, pregnancy and/or breast feeding, coagulopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with GIM under endoscopic surveillance or examination at Qilu Hospital from March 1 to September 31, 2015 were recruited into this study. 94 patients were eligible for analysis (50 males and 44 females; average age 53 years, range 22-80 years).
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
blood flow state | 5 months
  Flow determination cannot yet be done automatically. It requires a semi-quantitative analysis involving subjective assessment. Assessment of flow determination was based on the previously published consensus criteria, in which flow was classified into seven grades.
  Flow was categorized as: "linear flow" (fast and continuous flow, like plastic tape without grainy), "linear particle flow"(fast and continuous flow, like ribbon with mild grainy), "particle linear flow"(fast and continuous flow, like cotton tape with obvious grainy), "particle flow"(sluggish flow like mud-sand flow), "slowly particle flow"(slow but continuous), "particle of pendulum flow"(swinging silt flow) and "stagnate"(no flow).
microvascular area in μm2 | 5 months
  We analyzed the CLE images by using Adobe PhotoShop CS6 software. Ten images selected randomly and good displays of the vascular network were chosen from each sample for the analysis of the vascular structures. The Picture Cutout Guide and straight line tool were used to manually measure the area and length of each vascular segment. Each vascular segment was labeled and measured. We defined the microvascular length as the ratio of microvascular area to the microvascular diameter. The final measurement results of the microvascular area and diameter are the average of the 10 groups' testing values, respcetively. The results were exported in an Excel file and reported as the mean ± standard error (SD) for each individual case.
microvascular diameter in μm | 5 months
  We analyzed the CLE images by using Adobe PhotoShop CS6 software. Ten images selected randomly and good displays of the vascular network were chosen from each sample for the analysis of the vascular structures. The Picture Cutout Guide and straight line tool were used to manually measure the area and length of each vascular segment. Each vascular segment was labeled and measured. We defined the microvascular length as the ratio of microvascular area to the microvascular diameter. The final measurement results of the microvascular area and diameter are the average of the 10 groups' testing values, respcetively. The results were exported in an Excel file and reported as the mean ± standard error (SD) for each individual case.

SECONDARY OUTCOMES:
vascular morphology | 5 months
  It included normal or tortuous and dilation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China